CLINICAL TRIAL: NCT06489444
Title: Alterations in Nutrient-sensing Mechanisms May Play a Role in Symptom Generation in Patients With IBS
Brief Title: Fecal Amino Acids，Gut Taste Receptors and Irritable Bowel Syndromes
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital of Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023232
Record Dates: First submitted 2024-03-16; First posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- IBS-D
- IBS-C
- Health control
- UC(ulcerative colitis)

SUMMARY:
Clinical data, fresh feces and intestinal mucosal tissues of patients with diarrheal IBS were collected. High performance liquid chromatography, immunohistochemistry and immunofluorescence were used to study the amino acid levels in feces of patients with IBS, the expression of taste receptors in intestinal mucosa, and the correlation between symptoms of abdominal pain and diarrhea and the expression of taste receptors, so as to obtain the conclusion that "intestinal amino acid perception abnormalities exist in patients with IBS. And correlated with clinical symptoms."

ELIGIBILITY:
Inclusion Criteria:

* Patients with IBS who meet the Rome IV diagnostic criteria:

  1. that is, recurrent abdominal pain, with symptoms occurring at least 1 day per week or at least 3 days per month on average in the last 3 months, combining 2 or more of the following:

     1. related to defecation;
     2. accompanied by changes in the frequency of bowel movements;
     3. Accompanied by changes in fecal characteristics (appearance). (Symptoms appeared at least 6 months before diagnosis, and above diagnostic criteria were met in the last 3 months) 2. Age ≥18 years old.

Exclusion Criteria:

* 1. History of celiac disease and other organic intestinal diseases, metabolic diseases (thyroid dysfunction, diabetes, etc.); (2) Serious neurological, mental and psychological diseases, or accompanied by serious organ dysfunction; 3. Abdominal surgery; 4. Pregnant, possible pregnant and lactating patients; 5. History of colonoscopy in the past 1 year; 6. Declined to participate in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with irritable bowel syndrome who met all inclusion and exclusion criteria and corresponding healthy controls admitted to the gastroenterology Department of the Second Affiliated Hospital of Xi 'an Jiaotong University
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-03-16 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Taste receptor expression was associated with symptom severity | 1 year
  The severity of symptoms was correlated with the expression of taste receptors
Association between fecal amino acid levels and symptom severity in patients | 1year
  The severity of symptoms was correlated with fecal amino acid

CONTACTS AND LOCATIONS:
Locations (1):
- The second affiliated hospital of xi'an jiaotong university, Xi'an, Shaanxi, China